CLINICAL TRIAL: NCT06140615
Title: The Utility of Lung Ultrasound Scores to Determine Extubation Readiness in Neonates With Respiratory Distress on Mechanical Ventilation
Brief Title: Lung Ultrasound - Prospective Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Meriter Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-1751; 2023-026 (Other: Meriter); non-PBA dated 7/8/24 (Other: Meriter); 2023-1132 (Other: UW Madison)
Record Dates: First submitted 2023-11-14; First posted 2023-11-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Distress of Newborn
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lung ultrasound (Experimental): Participants undergo pre- and post-extubation lung ultrasound
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound of lungs

SUMMARY:
The goal of this clinical trial is to determine whether lung ultrasound can predict extubation success in neonates with respiratory distress.

Participants will undergo a lung ultrasound pre- and post-extubation.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at UnityPoint Health Meriter Hospital and University of Minnesota admitted to the Neonatal Intensive Care Unit (NICU) with respiratory distress requiring intubation
* Meeting the extubation readiness criteria per the attending neonatologist

Exclusion Criteria:

* Known major congenital disease (chromosomal abnormality, heart disease, respiratory malformation)
* Neonates with parents that are less than 18 years old

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Ability of lung ultrasound score to predict extubation success | 12 hours pre-extubation to 24 hours post extubation
  Correlate the lung ultrasound score to the success of extubation, which is defined as remaining extubated for >72 hours. Ultrasound scores are measured on a 4-point scale (0=normal,3 = most abnormal).

SECONDARY OUTCOMES:
Change in pre- and post-extubation lung ultrasound scores | 12 hours pre-extubation to 24 hours post extubation
  Ultrasound scores are measured on a 4-point scale (0=normal,3 = most abnormal).
Time to re-intubation | Up to 72 hours post-intubation
  Length of time from extubation to re-intubation.
Change in heart rate | 5 minutes before to 5 minutes after lung ultrasound
  Measure of heart rate before and after ultrasound procedure
Change in respiratory rate | 5 minutes before to 5 minutes after lung ultrasound
  Measure of respiratory rate before and after ultrasound procedure
Change in oxygen saturation | 5 minutes before to 5 minutes after lung ultrasound
  Measure of oxygen saturation before and after ultrasound procedure

CONTACTS AND LOCATIONS:
Overall Officials: Adam S Bauer, MD, Principal Investigator — Meriter Foundation
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Unity-Point Health Meriter, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No